CLINICAL TRIAL: NCT05033574
Title: The State of Sexual Development in Children With Inherited Epidermolysis Bullosa
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Medical Research Center for Children's Health, Russian Federation (Other Government)
Responsible Party: Sponsor
Other Study IDs: 6
Record Dates: First submitted 2021-07-25; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-07

CONDITIONS: Dermatologic Disease; Epidermolysis Bullosa; Epidermolysis Bullosa Simplex; Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa, Junctional; Kindler Syndrome; Puberty Disorders; Hormone Disturbance
Keywords: inherited epidermolisys bullosa; epidermolisys bullosa; epidermolisys bullosa simplex; epidermolisys bullosa junctional; epidermolisys bullosa dystrophic; Kindler syndrome; puberty; sexual development; epidermolysis bullosa; congenital epidermolysis bullosa
MeSH Terms: conditions — Skin Diseases; Epidermolysis Bullosa; Epidermolysis Bullosa Simplex; Epidermolysis Bullosa Dystrophica; Epidermolysis Bullosa, Junctional; Poikiloderma of Kindler; Endocrine System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Prepubescent and pubertal girls with an established diagnosis of epidermolysis bullosa simplex: Female patients aged 8 to 18 years with a diagnosis of epidermolysis bullosa simplex.
  Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist
- Prepubescent and pubertal girls with an established diagnosis of junctional epidermolysis bullosa: Female patients aged 8 to 18 years with a diagnosis of junctional epidermolysis bullosa.
  Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist
- Prepubescent and pubertal girls with an established diagnosis of epidermolysis bullosa dystrophic: Female patients aged 8 to 18 years with a diagnosis of epidermolysis bullosa dystrophic.
  Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist
- Prepubescent and pubertal girls with an established diagnosis of Kindler syndrome: Female patients aged 8 to 18 years with a diagnosis of Kindler syndrome. Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist
- Prepubescent and pubertal boys with an established diagnosis of epidermolysis bullosa simplex: Male patients aged 8 to 18 years with a diagnosis of epidermolysis bullosa simplex.
  Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist
- Prepubescent and pubertal boys with an established diagnosis of junctional epidermolysis bullosa: Male patients aged 8 to 18 years with a diagnosis of junctional epidermolysis bullosa.
  Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist
- Prepubescent and pubertal boys with an established diagnosis of epidermolysis bullosa dystrophic: Male patients aged 8 to 18 years with a diagnosis of epidermolysis bullosa dystrophic.
  Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist
- Prepubescent and pubertal boys with an established diagnosis of Kindler epidermolysis bullosa: Male patients aged 8 to 18 years with a diagnosis of Kindler syndrome. Based on the results of diagnostic methods, further division of patients into prepubertal and pubertal periods of puberty is planned.
  Interventions: Diagnostic Test: Biochemical study of hormone levels; Diagnostic Test: Ultrasound examination; Radiation: Radiography of the hands; Behavioral: Consultation of a medical psychologist

INTERVENTIONS:
Diagnostic Test: Biochemical study of hormone levels — Biochemical study of the level of follicle-stimulating hormone, luteinizing hormone, estradiol, total testosterone, prolactin, 17-hydroxyprogesterone, dehydroepiandrosterone sulfate, cortisol, insulin, thyroid-stimulating hormone, tetraiodothyronine, thyr
Diagnostic Test: Ultrasound examination — Ultrasound examination of the pelvic organs in girls and the scrotum organs in boys
Radiation: Radiography of the hands — Determination of bone age using radiography of the hands
Behavioral: Consultation of a medical psychologist — Consultation with a medical psychologist to determine the patient's psychological condition and level of intelligence

SUMMARY:
The aim of the study is to determine the state of sexual development in patients with inherited epidermolysis bullosa; the study is planned to include boys and girls aged 8 to 18 years with a diagnosis of epidermolysis bullosa simplex, junctional epidermolysis bullosa, Kindler syndrome.

DETAILED DESCRIPTION:
Determination of sexual development in children with various types of inherited epidermolysis bullosa using clinical, laboratory and instrumental methods for diagnosing the condition.

Phenotyping of patients with inherited epidermolysis bullosa, taking into account their physical and sexual development, indicators of self-attitude and socialization.

Development of algorithms for individual care for patients with inherited epidermolysis bullosa, including an assessment of the psychological state at different age stages (primary school and adolescence), the volume and form of psychological and pedagogical assistance in complex rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 8 to 18 years of age with an established diagnosis of epidermolysis bullosa simplex, junctional epidermolysis bullosa, dystrophic epidermolysis bullosa, Kindler syndrome.

Exclusion Criteria:

1. Hypergonadotropic hypogonadism;
2. previous treatment with sex steroids or gonadotropins;
3. the presence of endocrine diseases (hypothyroidism, hypercorticism, hyperprolactinemia, diabetes mellitus);
4. the presence of chronic somatic diseases that are not complications of inherited epidermolysis bullosa (bronchopulmonary diseases, cardiovascular diseases, diseases of the urinary system, diseases of the gastrointestinal tract).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female patients from 8 to 18 years of age with an established diagnosis of epidermolysis bullosa simplex, junctional epidermolysis bullosa, dystrophic epidermolysis bullosa, Kindler syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the state of sexual development of children with various types of inherited epidermolysis bullosa using the Tanner scale | 1 day
  The endocrinologist's assessment of pubertal development in boys and girls using the Tanner Scale
Determination of the state of functional activity of the sex glands in children with various types of inherited epidermplysis bullosa by the method of biochemical study of the level of sex hormones | 1 day
  Determination of serum levels of sex hormones in patients (luteinizing hormone, follicle-stimulating hormone, estradiol, total testosterone).
Determination of additional hormonal indicators | 1 day
  Determination of blood levels of adrenocorticotropic hormone, cortisol, dehydroepiandrosterone-sulfate, 17-hydroxyprogesterone, prolactin, insulin, thyrotropic hormone, triiodothyronine and thyroxine.
Functional development and morphometric parameters of the genital glands in children with various types of inherited epidermolysis bullosa by ultrasound diagnostics | 1 day
  Ultrasound examination of pelvic organs in girls and scrotal organs in boys to determine morphometric indices.
The state of bone age in children with various types of inherited epidermolysis bullosa using X-ray examination of the hands | 1 day
  Determination of bone and chronological age correspondence by radiography of the left wrist joint.
Determination of the psychological state of children with various types of inherited epidermolysis bullosa using the Pearce-Harris scale | 1 day
  Determination of the relationship between self-esteem and gender development in children with different types of hereditary epidermolysis bullosa using the Peirce-Harris scale
Determination of the psychological state of children with various types of inherited epidermolysis bullosa using the personality drawing technique of K. Machover | 1 day
  Determination of the relationship between self-esteem and gender development in children with different types of hereditary epidermolysis bullosa using the personality drawing technique of K. Machover
Determination of the psychological state of children with various types of inherited epidermolysis bullosa using the T. Aachenbach questionnaire | 1 day
  Determination of the relationship between self-esteem and gender development in children with different types of hereditary epidermolysis bullosa using the T. Aachenbach questionnaire
Determination of the level of intellectual development in children with various types of inherited epidermolysis bullosa using D. Wexler's test | 1 day
  Determination of the level of intellectual development and its components (verbal and non-verbal intelligence) in children with various types of inherited epidermolysis bullosa
Determination of the severity of the course of the disease in children with various types of inherited epidermolysis bullosa using EBDASI | 1 day
  Determination of the severity of the course of the disease in children with various types of inherited epidermolysis bullosa using Epidermolysis Bullosa Disease Activity and Scarring Index (EBDASI)

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical Research Center for Children's Health, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided